CLINICAL TRIAL: NCT00120471
Title: A Phase I Open Label Trial of the Safety and Pharmacokinetics of Tenofovir Disoproxil Fumarate in HIV-1 Infected Pregnant Women and Their Infants
Brief Title: Safety and Blood Levels of Tenofovir Disoproxil Fumarate in HIV Infected Pregnant Women and Their Babies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 057; 10143 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2005-07-14; First posted 2005-07-18 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Perinatal Transmission; MTCT; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

ARMS (4):
- 1 (Experimental): Pregnant participants will receive a single dose of TDF during active labor. These participants will be hospitalized at the delivery facility through Day 3 postpartum.
  Interventions: Drug: Tenofovir disoproxil fumarate
- 2 (Experimental): Pregnant participants will not receive TDF. Participants will be hospitalized at the delivery facility through Day 7 postpartum. Their infants will receive TDF at birth and on Days 3 and 5 after birth.
  Interventions: Drug: Tenofovir disoproxil fumarate
- 3 (Experimental): Pregnant participants will be hospitalized at the delivery facility through Day 7 postpartum. They will receive TDF during active labor and their infants will receive TDF at birth and on Days 3 and 5 after birth.
  Interventions: Drug: Tenofovir disoproxil fumarate
- 4 (Experimental): Pregnant participants will be hospitalized at the delivery facility through Day 7 postpartum. Mothers will receive TDF during active labor and their infants will receive TDF at birth and daily for 7 days after birth.
  Interventions: Drug: Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate — 600-mg tablet taken orally once daily
  Other Names: TDF
  Arms: 1; 3; 4
Drug: Tenofovir disoproxil fumarate — 4-mg/kg oral suspension taken at birth and on Days 3 and 5 after birth
  Other Names: TDF
  Arms: 2; 3
Drug: Tenofovir disoproxil fumarate — 6-mg/kg oral suspension taken at birth and daily for 7 days after birth
  Other Names: TDF
  Arms: 4

SUMMARY:
To prevent mother-to-child transmission (MTCT) of HIV in resource-limited countries, a simple yet effective treatment plan is needed. Tenofovir disoproxil fumarate (TDF) is an anti-HIV drug approved for use in the United States for the treatment of HIV infected adults. The purpose of this study is to determine the safety, tolerability, and blood levels of TDF in HIV infected pregnant women and their babies. The study will be conducted at sites in Malawi and Brazil.

DETAILED DESCRIPTION:
Rates of MTCT of HIV have dramatically decreased in resource-rich countries since the introduction of antiretroviral (ARV) prophylaxis; increased prenatal care, HIV testing, and counseling; elective cesarean delivery; and avoidance of breastfeeding. In resource-limited countries, however, MTCT of HIV continues to be a widespread problem. In these parts of the world, ARV prophylaxis is too expensive and too difficult to adequately administer; mothers often do not receive proper prenatal care; cesarean delivery may pose risks to the mother and and her infant; and due to the lack of safe, affordable, and socially acceptable alternatives, HIV infected mothers breastfeed their infants. The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of TDF in HIV infected pregnant women and their infants.

Participants in this study will be enrolled through 12 months after delivery. During the last trimester of pregnancy, HIV infected women will be screened for eligibility. Women will be enrolled into the study upon presentation at the study site for delivery. Standard of care with ARVs for prevention of MTCT will be offered to all women and their infants both inside and outside of the study; however, such ARVs will not be provided by this study.

There will be four cohorts in this study:

* Cohort 1 women will receive a single dose of TDF (SD TDF) during active labor. Cohort 1 women will be hospitalized at the delivery facility through Day 3 postpartum.
* Cohort 2 women will not receive any TDF. Cohort 2 women will be hospitalized at the delivery facility through Day 7 postpartum. Their infants will receive TDF at birth and on Days 3 and 5 after birth.
* Cohort 3 will not begin enrolling women until data safety evaluations of Cohorts 1 and 2 are completed. Cohort 3 women will be hospitalized at the delivery facility through Day 7 postpartum. Women in Cohort 3 will receive SD TDF during active labor, and their infants will receive TDF at birth and on Days 3 and 5 after birth.
* Cohort 4, which was added to the study based on a review of data from the other cohorts, will be similar to Cohort 3, except that infants will receive daily TDF for the 7 days after birth. Researchers believe this higher and more frequent dosing of TDF in infants will help them meet the target TDF concentration specified in the protocol.

There will be seven study visits for women at study entry (Day 0), Day 2, between Days 5 and 7, at Weeks 6 and 12, and at Months 6 and 12 postpartum. Medical history, a short physical exam, and blood collection will occur at all visits. In Cohorts 1, 3, and 4, blood collection for PK studies will occur prior to receiving TDF and seven times post-dose.

There will be eight study visits for infants, which will occur within 24 hours of birth; on Day 3; between Days 5 and 7; at Weeks 6 and 12; and at Months 6, 9, and 12. Medical history, a physical exam, and blood collection will occur at all visits. Infants will have x-rays to assess bone health at Day 3 and Month 3, except in Cohort 4, which will not include x-rays of infants. Infants of Cohort 1 will have blood collection for PK studies at birth and four times after birth. Infants of Cohorts 2 and 3 will undergo blood collections for PK studies at birth, Day 3, and Day 5. Blood collection at these visits will occur before receiving TDF and 2 and 10 hours after receiving TDF. At birth, an additional collection will occur 18 to 24 hours after receiving TDF, and on Day 5, two additional collections will occur--at 18 to 24 hours and at 36 to 48 hours after receiving TDF. Infants of Cohort 4 will have blood collection for PK studies at birth and after their fourth and seventh doses of TDF.

ELIGIBILITY:
Inclusion Criteria for HIV Infected Pregnant Women:

* HIV-1 infected
* Intend to deliver at the study site
* Willing to be contacted or visited at home
* Willing to be admitted to and remain in the delivery facility through Day 3 postpartum (Cohort 1) or Day 7 postpartum (Cohorts 2 and 3)

Exclusion Criteria for HIV Infected Pregnant Women:

* Prior treatment with TDF
* Active opportunistic infection
* Serious bacterial infection
* Chronic malabsorption or diarrhea during the current pregnancy
* Clinically significant disease or condition that, in the opinion of the study clinician, would interfere with the study
* Known multiple gestation (twins, etc.) prior to study entry
* Participation in any other therapeutic or vaccine trial during the current pregnancy
* Use of certain medications
* Any other condition or situation that, in the opinion of the investigator, would interfere with the study
* For Cohort 4, use of atazanavir or lopinavir/ritonavir (Kaletra) within 2 weeks of anticipated delivery

Exclusion Criteria for Infants Born to HIV Infected Pregnant Women:

* Birth weight of less than 2 kg (4.4 lbs)
* Severe congenital malformation or other medical condition that may affect survival and, in the opinion of the clinician, participation in this study
* Grade 2 or higher serum creatinine level or any other Grade 3 or higher toxicity
* Part of a multiple birth (twins, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2006-11; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events with a severity of Grade 3 or higher attributable to receipt of TDF | Throughout study
Maintenance of infant serum concentrations of TDF greater than 50 ng/ml | Through Week 1

SECONDARY OUTCOMES:
Maternal HIV-1 RNA levels | At study entry, Days 5 to 7, and Week 6
Viral resistance to TDF in all HIV-1 infected infants, all of the corresponding mothers (transmitters), and a subset of mothers whose infants are not infected (nontransmitters). Analysis of TDF in mothers may include testing of breastmilk samples. | Throughout study
HIV infection in infants | Throughout study
TDF concentration in amniotic fluid and breast milk | Through Week 1

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mirochnick, MD, Study Chair — Boston Medical Center; Taha Taha, MD, PhD, Study Chair — Johns Hopkins University; Regis Kreitchmann, MD, Study Chair — Centro Municipal de DST/AIDS, Irmandade Santa Casa de Misericordia de Porto Alegre
Locations (5):
- Brazil (4):
  - Federal Univ. of Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital Nossa Senhora da Conceicao CRS, Porto Alegre, Rio Grande do Sul
  - Irmandade Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - HSE-Hospital dos Servidores do Estado CRS, Rio de Janeiro
- College of Med. JHU CRS, Blantyre, Malawi

REFERENCES:
- [Background] Abrams EJ. Prevention of mother-to-child transmission of HIV--successes, controversies and critical questions. AIDS Rev. 2004 Jul-Sep;6(3):131-43. PMID 15595430
- [Background] Capparelli E, Rakhmanina N, Mirochnick M. Pharmacotherapy of perinatal HIV. Semin Fetal Neonatal Med. 2005 Apr;10(2):161-75. doi: 10.1016/j.siny.2004.10.001. Epub 2005 Jan 20. PMID 15701581
- [Background] Thorne C, Newell ML. Mother-to-child transmission of HIV infection and its prevention. Curr HIV Res. 2003 Oct;1(4):447-62. doi: 10.2174/1570162033485140. PMID 15049430
- [Background] Capparelli EV, Englund JA, Connor JD, Spector SA, McKinney RE, Palumbo P, Baker CJ. Population pharmacokinetics and pharmacodynamics of zidovudine in HIV-infected infants and children. J Clin Pharmacol. 2003 Feb;43(2):133-40. doi: 10.1177/0091270002239821. PMID 12616665
- [Derived] Osorio LE, Boechat MI, Mirochnick M, Kumwenda N, Kreitchmann R, Emel L, Pinto J, Joao E, Santos B, Swenson M, George K, Sato P, Mofenson L, Nielsen-Saines K; HIV Prevention Trials Network (HPTN) 057 Protocol Team. Bone Age and Mineral Density Assessments Using Plain Roentgenograms in Tenofovir-exposed Infants in Malawi and Brazil Enrolled in HIV Prevention Trials Network 057. Pediatr Infect Dis J. 2017 Feb;36(2):184-188. doi: 10.1097/INF.0000000000001386. PMID 27798550